CLINICAL TRIAL: NCT04245605
Title: Invasive Coronary Angiography Early in Ischemic Heart Failure (ICE-HF)
Brief Title: Invasive Coronary Angiography Early in Ischemic Heart Failure
Acronym: ICE-HF
Status: Completed | Type: Observational
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Douglas Lee, Principal Investigator, Institute for Clinical Evaluative Sciences
Other Study IDs: 3
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Acute Heart Failure
Keywords: Coronary angiography; Invasive strategy; Myocardial infarction; Troponin; Heart failure
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early angiography: Patients admitted to hospital with acute heart failure undergoing coronary angiography within 14 days of hospital admission
  Interventions: Procedure: Coronary angiography
- Control: Patients admitted to hospital with acute heart failure not undergoing coronary angiography within 14 days

INTERVENTIONS:
Procedure: Coronary angiography — Coronary angiogram performed either in hospital or post-discharge, within 14 days after initial hospital presentation with heart failure
  Other Names: Diagnostic coronary angiography
  Groups: Early angiography

SUMMARY:
To compare the outcomes of patients with acute heart failure who undergo early coronary angiography vs. usual care

ELIGIBILITY:
Inclusion Criteria: Adult patients with acute heart failure, hospitalized in Ontario, Canada, with evidence of possible ischemic heart disease, defined as at least one of: a) prior myocardial infarction, b) troponin elevation, or c) angina.

Exclusion Criteria:

* Recent myocardial infarction
* Coronary angiogram or revascularization within previous 3 months before admission
* Nonresidents of Ontario, invalid health card number
* HF diagnosed after admission
* Admission BNP or NT-proBNP not diagnostic of HF
* Died within 14 days of admission
* Palliative within 6 months prior to hospital admission
* Elevated creatinine concentration
* Documented anaphylactic contrast allergy
* Ischemic or hemorrhagic stroke within 3 months prior to admission
* Highest category of Hospital Frailty Risk Score
* Active severe bleeding at time of hospital admission
* Absolute platelet count < 20
* Metastatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-described male or female
Study Population: Hospitalized patients in Ontario, Canada with acute heart failure
Sampling Method: Probability Sample
Enrollment: 2994 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 2 years
  Death from any cause after 14 days in landmark analysis
Cardiovascular mortality | 2 years
  Death due to cardiovascular causes after 14 days in landmark analysis

SECONDARY OUTCOMES:
All-cause hospital readmission | 2 years
  Readmissions for all causes after 14 days or hospital discharge in landmark analysis
Heart failure readmission | 2 years
  Readmissions for heart failure after 14 days or hospital discharge in landmark analysis
Readmission for myocardial infarction | 2 years
  Readmissions for myocardial infarction after 14 days or hospital discharge in landmark analysis
Rates of revascularization | 90 days
  Coronary revascularization with CABG surgery or PCI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Lee, MD, PhD, Principal Investigator — ICES
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No